CLINICAL TRIAL: NCT00726804
Title: Discontinuation of TNF-alpha Inhibitors in Spondylarthritis Patients With Low Disease Activity, and Re-initiation of Therapy if Disease Flares
Brief Title: Discontinuation of TNF-alpha Inhibitors in Patients With Spondyloarthritis
Acronym: SPARTA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: It was not possible to recruit patients
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, MOstergaard, Professor, Glostrup University Hospital, Copenhagen
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPARTA
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: SPONDYLOARTHRITIS
MeSH Terms: conditions — Spondylarthritis | interventions — Etanercept; Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2 (Other)
  Interventions: Drug: Discontinuation of TNF-alpha inhibitor and re-starting it if flare-up in disease activity (etanercept or adalimumab)

INTERVENTIONS:
Drug: Discontinuation of TNF-alpha inhibitor and re-starting it if flare-up in disease activity (etanercept or adalimumab) — Discontinuation of infusion infliximab (Remicade) 3-5mg/kg every 6-8 week, injection of etanercept (Enbrel) 25 mg x 2/week or injection of adalimumab (Humira) 40 mg eow.

SUMMARY:
Spondylarthropathy (SpA) comprises a group of rheumatic diseases mainly affecting the spine and sacroiliac joints. In most of the patients disease activity alternates, and some patients have symptom free periods. Tumor-Necrosis-Factor-alpha (TNF-alpha) antagonists have significantly improved the treatment options for patients with spondyloarthritis. TNF-alpha antagonist therapy is costly, implies an increased risk of infections, including reactivation of tuberculosis, and the risk of long-term adverse events, as cancer, is fully clarified. It is highly relevant to explore to which extent anti-TNF-alpha therapy can be discontinued in SpA patients without immediate relapse of disease activity. Two studies have investigated discontinuation of a TNF-alpha antagonist (infliximab and etanercept) in ankylosing spondylitis, reporting flares in the majority of patients within the 1-year follow-up period, with the longest times to relapse in patients with the lowest disease activity. The effect of adalimumab discontinuation has never been studied, and, furthermore, the effect of TNF-alpha-antagonist discontinuation has never been studied in patients with early spondyloarthritis not fulfilling the New York criteria.

ELIGIBILITY:
Inclusion Criteria:

1. At least 12 months of treatment with infliximab, etanercept and adalimumab.
2. Diagnosis of spondylarthritis according to the European Spondyloarthritis Study Group (ESSG) criteria or modified New York Criteria
3. No clinical active disease, defined as a BASDAI score < 4.
4. Among other issues: Age >18 years; written informed consent, adequate birth control; no contraindications for anti-TNF-alpha-therapy

Exclusion Criteria:

1. Treatment with disease modifying anti-rheumatic drugs within 4 weeks before screening
2. Oral, intraarticular, intramuscular or intravenous glucocorticoid within 4 weeks before screening
3. Pregnancy or lactation
4. HIV, hepatitis B or C, tuberculosis, other infections
5. Malignancies
6. Other serious concomitant diseases (uncontrolled/severe kidney, liver, haematological, gastrointestinal, endocrine, cardiovascular, pulmonary, neurological ore cerebral disease (including demyelinating disease)
7. Contraindications to anti-TNF-alpha-therapy
8. Contraindications to MRI

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Flair-up in disease activity in axial arthritis and therapeutic response at re-starting TNF-alpha inhibitors | 40 weeks

SECONDARY OUTCOMES:
Bath ankylosing spondylitis disaease activity score, Bath ankylosing spondylitis functional index, Bath ankylosing spondylitis metrology index, C-Reactive protein, MRI, biomarkers of inflammation, cartilage and bone turnover | 40 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel Østergaard, Professor, Study Chair — Department of rheumatology, Glostrup Hospital, Copenhagen; Susanne J Pedersen, MD, Study Chair — Department of rheumatology, Glostrup Hospital, Copenhagen; Inge J Sørensen, MD, PhD, Study Chair — Department of rheumatology, Glostrup Hospital, Copenhagen
Locations (4):
- Denmark (4):
  - Glostrup Hospital, Copenhagen
  - Gentofte Hospital, Copenhagen
  - Gråsten Gigthospital, Gråsten
  - Vejle Sygehus, Vejle